CLINICAL TRIAL: NCT03344185
Title: The Effect of Glycaemic Index Variation on Blood Glucose and Mood in Healthy Participants Across the Day
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Matthew Grout (Other)
Responsible Party: Sponsor-Investigator, Matthew Grout, Doctoral Researcher, University of Reading
Organization: University of Reading (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2016-032-DL
Record Dates: First submitted 2017-11-09; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Mood; Diet Modification; Glucose, Low Blood; Glucose, High Blood
Keywords: glycaemic index; mood; glucose; diet

STUDY DESIGN:
Intervention Model Description: All participants took part in both diet conditions
Who Masked: Participant
Masking Description: Participants were not told which diet they were consuming each day.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low GI diet (Experimental): This diet contained three meals, all with a low GI value. This was the Low Glycaemic Diet intervention.
  Interventions: Dietary Supplement: Low Glycaemic Diet
- High GI diet (Experimental): This diet contained three meals, all with a high GI value. This was the High Glycaemic Diet intervention.
  Interventions: Dietary Supplement: High Glycaemic Diet

INTERVENTIONS:
Dietary Supplement: Low Glycaemic Diet — This intervention consisted of three low GI meals.
  Arms: Low GI diet
Dietary Supplement: High Glycaemic Diet — This intervention consisted of three meals, all with a high GI value.
  Arms: High GI diet

SUMMARY:
This study provided 24 healthy subjects with two diets that varied in their glycaemic index values. One condition was a low GI diet, whilst the other was a high GI diet. Glucose concentrations and mood were measured throughout each test day.

DETAILED DESCRIPTION:
Therefore, the aim of this study is to feed to participants meals which differing in their glycaemic index across the course of a day, and thus produce different glycaemic responses. The outcome variables will be blood glucose levels and subjective mood. The purpose of this study is to identify the appropriate times (according to glycaemic response) at which cognitive functioning should be tested. Importantly, this study is also the first step to characterizing glycaemic and cognitive profiles associated with food consumption over a whole day (breakfast, lunch, snack) rather than just one meal (e.g. breakfast), ranging from the most favourable (stable glucose regulation) to the least favourable (variability; many peaks and troughs).

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years of age.
* Willing to participate in the entire study (signed informed consent required)
* Subjects will be eligible for the study if male or female (not pregnant or lactating)

Exclusion Criteria:

* Diabetic
* Smoker
* Have any food intolerances or allergies
* History of alcohol or drug misuse
* Diagnosed with any of the following:

  * High blood cholesterol
  * High blood pressure
  * Thyroid disorder
  * Heart problems, stroke or any vascular disease in the past 12 months
  * Inflammatory diseases such as rheumatoid arthritis
  * Bone related conditions, such as osteoporosis
  * Renal, gastrointestinal, respiratory, liver disease or cancer
* You are presently taking part in another clinical trial or research study
* You are an elite athlete (very high intensity training more than 3 times a week)
* You are currently on a specific diet or taking any dietary supplements and are unwilling to cease during the testing period
* You are intending to regularly use medication which affects gastrointestinal motility

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in Glycaemic profile across the day | Assessed at 0 (baseline), 15, 30, 45, 60, 90, 120 mins after each meal. With 3 meals in a day this totaled 21 assessment point for each day, giving 42 assessment points to compare overall. Data will be reported for the duration of this 3 year PhD award.
  Change in blood glucose concentrations (mmol/L)

SECONDARY OUTCOMES:
Mood (alertness, anxiety and contentment) measured by Bond & Lader (1974) Visual Analogue Scale | This was measured 6 times a day (every 90 minutes starting at 0 minutes/baseline), giving a total of 12 times. Each time last approximately 5 minutes, giving a total of 60 minutes overall. Data will be reported for the duration of this 3 year PhD award.
  The Bond & Lader VAS provides participants with 16 lines measuring 100mm each. At the ends of each line are two words opposite in meaning. For example, 'alert' and 'drowsy'. A participants marks on the line closer to the word they currently feel. The score from each line is out of 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Lamport, PhD, Principal Investigator — University of Reading

IPD SHARING:
Plan to Share IPD: No